CLINICAL TRIAL: NCT03667651
Title: THE PEBBLES STUDY: A Randomised Controlled Trial to Prevent Eczema, Food Allergy and Sensitisation Using a Skin Barrier Improvement Strategy
Brief Title: The PEBBLES Study - Testing a Strategy for Preventing Eczema and Food Allergy in High Risk Infants
Acronym: PEBBLES
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Melbourne (Other)
Responsible Party: Principal Investigator, Adrian Lowe, Dr Adrian Lowe, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HREC/17/RCHM/221; ACTRN12617001380381 (Registry Identifier: Australian New Zealand Clinical Trials Registry)
Record Dates: First submitted 2018-09-09; First posted 2018-09-12 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Eczema; Asthma; Allergy;Food
MeSH Terms: conditions — Eczema; Asthma; Food Hypersensitivity | interventions — EpiCeram

STUDY DESIGN:
Intervention Model Description: A single blinded study design will be used
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to the group of allocation and will have no contact with the participants aside from the assessment of outcomes at six-weeks and 12-months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Twice daily use treatment with EpiCeram (Active Comparator): They will be instructed to apply EpiCeram™ to the full skin surface of their child twice per day for 6 months. The prophylactic use of EpiCeram™ is the intervention that is being tested for its effect on infant skin barrier function. We will instruct parents to apply approximately 6 grams of EpiCeram™ per application at two regular times each day, including after bathing the infant, or at the time they would normally bathe their child.
  Interventions: Drug: EpiCeram
- Standard skin care (No Intervention): Parents are to follow standard skin care practices

INTERVENTIONS:
Drug: EpiCeram — Parents will be instructed to apply EpiCeram™ to the full skin surface of their child twice per day for six months.
  Arms: Twice daily use treatment with EpiCeram

SUMMARY:
This is a phase III, single blind (outcome assessor is blinded), randomised controlled multicentre trial of the effect of EpiCeram emollient for improving and maintaining skin barrier function and reducing incidence of eczema and food allergy in high risk infants.

A total of 760 participants with a first degree family history of allergic disease (asthma, eczema, allergic rhinitis or food allergy) will be recruited (380 each group) from maternity wards of three hospitals.

DETAILED DESCRIPTION:
The primary objective of this study is to demonstrate that twice daily application of a ceramide dominant emollient reduces the risk of eczema and food allergy, when compared to standard skin management. Secondary objectives are to determine if twice daily application of a ceramide dominant emollient reduces the risk of infants developing allergic sensitisation (as measured by skin prick test); to determine if twice daily application of a ceramide dominant emollient improves infant skin barrier function; to determine the level of parental compliance with a program to build infant skin barrier function; to confirm that a ceramide dominant emollient does not cause adverse effects in infants; to determine the level of compliance required to demonstrate an improvement in infant skin barrier function and to determine if twice daily application of a ceramide dominant emollient influences infant skin microbial colonisation, or skin lipid profile.

This is a phase III, single blind (outcome assessor is blinded), randomised controlled multicentre trial of the effect of EpiCeram emollient for improving and maintaining skin barrier function and reducing incidence of eczema and food allergy in high risk infants.

A total of 760 participants with a first degree family history of allergic disease (asthma, eczema, allergic rhinitis or food allergy) will be recruited (380 each group) from maternity wards of three hospitals.

Treatment will be from birth until six months, with a six week, six month and twelve month follow-up. An initial assessment will be performed at baseline which incorporates three surveys, a skin assessment, diary card (which is to be completed weekly and measures compliance), a breast milk sample, guthrie card and tape stripping. The six week and six month assessments entail a skin assessment, survey, compliance check, breast milk sample, tape stripping and guthrie card. Primary outcomes are assessed at the 12 month follow up where in addition to the aforementioned items, a saliva sample will also be taken and skin prick testing and food challenges will be performed when children have a positive SPT to one or more foods..

ELIGIBILITY:
Inclusion Criteria:

Infants will be eligible for this study if their mother, father, or an older sibling has a self-reported history of at least one of the following conditions:

* asthma,
* eczema/atopic dermatitis,
* hay fever/ allergic rhinitis or
* food allergy

Exclusion Criteria: infants with any of the following will be excluded:

* A parent who has a known hypersensitivity to any of the ingredients of EpiCeram™ will be excluded, as it would be difficult for these parents to apply EpiCeram™ to their infant, and there is likely to be an increased risk of the infant reacting to the cream.
* Multiple births (twins, triplets etc.) will be excluded, due to the difficulty in randomising individual twins and because of the clustering effect of multiple children from the same family which would reduce the effective sample size of the study.
* Who are born premature (<36 weeks) as the effect of the intervention may be different in premature infants.
* Who have major birth or early life medical complications that require admission into a special care nursery, as it will be difficult for parents to comply with the study requirements.
* Whose parents do not have sufficient English language skills to be able to answer questions.
* Whose parents are not able to comply with all protocol required visits and procedures

Max Age: 3 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 760 (Estimated)
Dates: Start 2018-03-06 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Presence of eczema | 12 months of age.
  as assessed using i) the UK working party criteria for eczema and/or ii) blinded investigator observed eczema.
Confirmed diagnosis of food allergy at 12 months (52 weeks). | 12 months of age
  This diagnosis is derived from a combination of allergic sensitisation, reaction history and food challenge. A skin prick test to six common allergens will be performed (egg white, cows' milk, peanut, dust mite, cat dander, and rye grass) along with a negative (saline) and a positive (histamine) control. Participants that are sensitised to certain foods (>=1mm wheal) during the skin prick testing will be given a challenge to determine if they are allergic to those foods. This will be conducted at the MCRI Allergy Clinic under the supervision of a Doctor specifically trained in oral food challenges.

SECONDARY OUTCOMES:
Eczema severity | 12 months of age
  assessed using the EASI score
Parent report of a community doctor diagnosis of eczema | 12 months of age
infant skin barrier function | At 6 weeks and 12 months of age
  As assessed by Trans-epidermal water loss (Vapometer)
Parental compliance with a program to build infant skin barrier function | At 6 weeks and 6 months of age.
  as assessed by parental completion of weekly diary cards and weighing of the tubes of study cream at each visit
Adverse events | From recruitment of infant until final study visit at 12 months of age.
  as assessed by the documentation of any untoward medical occurrence in a participant enrolled into this study
skin microbial colonisation, or skin lipid profile | At 6 weeks and 6 and 12 months of age
  Assessed using skin swabs at baseline, 6 weeks and 12 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Adrian J Lowe, Doctorate, Principal Investigator — University of Melbourne
Locations (4):
- Australia (4):
  - Mercy Women's Hospital, Heidelberg, Victoria
  - Frances Perry Private Hospital, Parkville, Victoria
  - Murdoch Children's Research Institute, Parkville, Victoria
  - Royal Women's Hospital, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lowe A, Su J, Tang M, Lodge CJ, Matheson M, Allen KJ, Varigos G, Sasi A, Cranswick N, Hamilton S, Robertson CF, Hui J, Abramson M, O'Brien S, Dharmage S. PEBBLES study protocol: a randomised controlled trial to prevent atopic dermatitis, food allergy and sensitisation in infants with a family history of allergic disease using a skin barrier improvement strategy. BMJ Open. 2019 Mar 13;9(3):e024594. doi: 10.1136/bmjopen-2018-024594. PMID 30867201